CLINICAL TRIAL: NCT05962008
Title: Effects of Consumption of Phosphatidylserine on the Cognitive Function: a Randomized, Placebo-controlled, Double-blind, Parallel-group Comparison Study
Brief Title: Effects of Consumption of Phosphatidylserine on the Cognitive Function
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Orthomedico Inc. (Other)
Collaborators: ECA Healthcare Inc. (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 06788-0019-10
Record Dates: First submitted 2023-07-04; First posted 2023-07-27 (Actual); Last update posted 2024-08-02 (Actual); Status verified 2024-08

CONDITIONS: Healthy Japanese Subjects
Keywords: Phosphatidylserine; Cognitive function

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Omega-3-phosphatidylserine derived from herring roe (Active Comparator): Take 300 mg/day of omega-3-phosphatidylserine derived from herring roe.
  Interventions: Dietary Supplement: DHAPS® product
- Phosphatidylserine derived from soybean (Active Comparator): Take 300 mg/day of phosphatidylserine derived from soybean.
  Interventions: Dietary Supplement: BioPS® product
- Placebo (Placebo Comparator): Take 0 mg/day of phosphatidylserine.
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: DHAPS® product — Take 4 capsules per day after breakfast with warm water.
  Arms: Omega-3-phosphatidylserine derived from herring roe
Dietary Supplement: BioPS® product — Take 4 capsules per day after breakfast with warm water.
  Arms: Phosphatidylserine derived from soybean
Dietary Supplement: Placebo — Take 4 capsules per day after breakfast with warm water.
  Arms: Placebo

SUMMARY:
The main objective of this trial is to verify the effects of consumption of phosphatidylserine for 12 weeks on the cognitive function in healthy Japanese subjects.

DETAILED DESCRIPTION:
In this study, the investigators will evaluate the cognitive function before and after the intervention. The groups to be compared are omega-3-phosphatidylserine derived from herring roe, phosphatidylserine derived from soybean, and a placebo.

ELIGIBILITY:
Inclusion Criteria:

1. Japanese
2. Male and female
3. Subjects aged 35-65
4. Healthy subjects
5. Subjects who notice a decline in memory
6. Subjects whose scoring of Mini Mental State Examination (MMSE) is 24 or more
7. Subjects who met the inclusion criteria 1. ~ 6. and have relatively low standardized score in composite memory measured using Cognitrax at Scr (Selection of those with relatively low standardized scores will be conducted in blocks of "Subjects aged 50 or over" and "Subjects aged under 50")
8. Subjects who are judged as eligible to participate in the study by the physician

Exclusion Criteria:

1. Subjects undergoing medical treatment or having a medical history of malignant tumor, heart failure, or myocardial infarction
2. Subjects carrying a pacemaker or an implantable cardioverter defibrillator (ICD)
3. Subjects undergoing treatment for any of the following chronic diseases: cardiac arrhythmia, liver disease, kidney disease, cerebrovascular disorder, rheumatism, diabetes mellitus, dyslipidemia, hypertension, or any other chronic diseases
4. Subjects who have dementia
5. Subjects who have mental health issues such as depression disorder, attention deficit/hyperactivity disorder (ADHD), or other issues
6. Subjects who use or take "Foods for Specified Health Uses", "Foods with Function Claims", or other functional food/beverage, as part of their daily intake
7. Subjects who take supplements or foods that may improve cognitive functions, such as phosphatidylserine, docosahexaenoic acid (DHA), eicosapentaenoic acid (EPA), ginkgo leaf extract, tocotrienol, astaxanthin, gamma-aminobutyric acid (GABA), and plasmalogen, as part of their daily intake
8. Subjects who take blue-backed fish such as sardines, mackerel, and saury for 4 days/week or over
9. Subjects who use devices, equipment, and applications that may affect cognitive functions (e.g., brain training puzzles, brain training games) as part of their daily life
10. Subjects regularly taking medications (including herbal medicines) and supplements
11. Subjects who are allergic to medications and/or the test food related products
12. Subjects who are pregnant, breast-feeding or planning for pregnancy during the trial period
13. Subjects who have been enrolled in other clinical trials 28 days before the agreement to participate in this trial or those who plan to enroll in another clinical trial during the trial period
14. Subjects who are deemed ineligible to participate by the principal investigator

Ages: 35 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 114 (Actual)
Dates: Start 2023-07-20 (Actual); Primary Completion 2024-03-17 (Actual); Study Completion 2024-03-17 (Actual)

PRIMARY OUTCOMES:
The measured value of the standardized score of composite memory at Week 12 | Week 12
  Verbal Memory (VBM) test and Visual Memory (VIM) test are measured using Cognitrax® which is powered by CNS Vital Signs®, a neurocognitive test system. The standardized score of composite memory is calculated from results of these two tests. This score has been normalized with a mean of 100 and a standard deviation of 15 based on age-matched reference data. Higher scores are always better.

SECONDARY OUTCOMES:
The amount of change of the standardized score of composite memory between Base line and Week 12 | Base line and Week 12
  VBM test and VIM test are measured using Cognitrax® which is powered by CNS Vital Signs®, a neurocognitive test system. The standardized score of composite memory is calculated from results of these two tests. This score has been normalized with a mean of 100 and a standard deviation of 15 based on age-matched reference data. Higher scores are always better.
The measured value of the standardized score of neurocognition index (NCI) at Week 12 | Week 12
  Seven neurocognitive tests {VBM, VIM, Finger Tapping (FTT), Symbol Digit Coding (SDC), Stroop Test (ST), Shifting Attention (SAT), and Continuous Performance (CPT)} are measured using Cognitrax® which is powered by CNS Vital Signs®, a neurocognitive test system. The standardized score of NCI is calculated from results of these seven tests. This score has been normalized with a mean of 100 and a standard deviation of 15 based on age-matched reference data. Higher scores are always better.
The amount of change of the standardized score of NCI between Base line and Week 12 | Base line and Week 12
  Seven neurocognitive tests {VBM, VIM, FTT, SDC, ST, SAT, and CPT} are measured using Cognitrax® which is powered by CNS Vital Signs®, a neurocognitive test system. The standardized score of NCI is calculated from results of these seven tests. This score has been normalized with a mean of 100 and a standard deviation of 15 based on age-matched reference data. Higher scores are always better.
The measured value of the standardized score of verbal memory at Week 12 | Week 12
  VBM test is measured using Cognitrax® which is powered by CNS Vital Signs®, a neurocognitive test system. The standardized score of verbal memory is calculated from the result of this test. This score has been normalized with a mean of 100 and a standard deviation of 15 based on age-matched reference data. Higher scores are always better.
The amount of change of the standardized score of verbal memory between Base line and Week 12 | Base line and Week 12
  VBM test is measured using Cognitrax® which is powered by CNS Vital Signs®, a neurocognitive test system. The standardized score of verbal memory is calculated from the result of this test. This score has been normalized with a mean of 100 and a standard deviation of 15 based on age-matched reference data. Higher scores are always better.
The measured value of the standardized score of visual memory at Week 12 | Week 12
  VIM test is measured using Cognitrax® which is powered by CNS Vital Signs®, a neurocognitive test system. The standardized score of visual memory is calculated from the result of this test. This score has been normalized with a mean of 100 and a standard deviation of 15 based on age-matched reference data. Higher scores are always better.
The amount of change of the standardized score of visual memory between Base line and Week 12 | Base line and Week 12
  VIM test is measured using Cognitrax® which is powered by CNS Vital Signs®, a neurocognitive test system. The standardized score of visual memory is calculated from the result of this test. This score has been normalized with a mean of 100 and a standard deviation of 15 based on age-matched reference data. Higher scores are always better.
The measured value of the standardized score of psychomotor speed at Week 12 | Week 12
  FTT test and SDC test are measured using Cognitrax® which is powered by CNS Vital Signs®, a neurocognitive test system. The standardized score of psychomotor speed is calculated from results of these two tests. This score has been normalized with a mean of 100 and a standard deviation of 15 based on age-matched reference data. Higher scores are always better.
The amount of change of the standardized score of psychomotor speed between Base line and Week 12 | Base line and Week 12
  FTT test and SDC test are measured using Cognitrax® which is powered by CNS Vital Signs®, a neurocognitive test system. The standardized score of psychomotor speed is calculated from results of these two tests. This score has been normalized with a mean of 100 and a standard deviation of 15 based on age-matched reference data. Higher scores are always better.
The measured value of the standardized score of reaction time at Week 12 | Week 12
  ST test is measured using Cognitrax® which is powered by CNS Vital Signs®, a neurocognitive test system. The standardized score of reaction time is calculated from the result of this test. This score has been normalized with a mean of 100 and a standard deviation of 15 based on age-matched reference data. Higher scores are always better.
The amount of change of the standardized score of reaction time between Base line and Week 12 | Base line and Week 12
  ST test is measured using Cognitrax® which is powered by CNS Vital Signs®, a neurocognitive test system. The standardized score of reaction time is calculated from the result of this test. This score has been normalized with a mean of 100 and a standard deviation of 15 based on age-matched reference data. Higher scores are always better.
The measured value of the standardized score of complex attention at Week 12 | Week 12
  ST test, SAT test, and CPT test are measured using Cognitrax® which is powered by CNS Vital Signs®, a neurocognitive test system. The standardized score of complex attention is calculated from results of these three tests. This score has been normalized with a mean of 100 and a standard deviation of 15 based on age-matched reference data. Higher scores are always better.
The amount of change of the standardized score of complex attention between Base line and Week 12 | Base line and Week 12
  ST test, SAT test, and CPT test are measured using Cognitrax® which is powered by CNS Vital Signs®, a neurocognitive test system. The standardized score of complex attention is calculated from results of these three tests. This score has been normalized with a mean of 100 and a standard deviation of 15 based on age-matched reference data. Higher scores are always better.
The measured value of the standardized score of cognitive flexibility at Week 12 | Week 12
  ST test and SAT test are measured using Cognitrax® which is powered by CNS Vital Signs®, a neurocognitive test system. The standardized score of cognitive flexibility is calculated from results of these two tests. This score has been normalized with a mean of 100 and a standard deviation of 15 based on age-matched reference data. Higher scores are always better.
The amount of change of the standardized score of cognitive flexibility between Base line and Week 12 | Base line and Week 12
  ST test and SAT test are measured using Cognitrax® which is powered by CNS Vital Signs®, a neurocognitive test system. The standardized score of cognitive flexibility is calculated from results of these two tests. This score has been normalized with a mean of 100 and a standard deviation of 15 based on age-matched reference data. Higher scores are always better.
The measured value of the standardized score of processing speed at Week 12 | Week 12
  SDC test is measured using Cognitrax® which is powered by CNS Vital Signs®, a neurocognitive test system. The standardized score of processing speed is calculated from the result of this test. This score has been normalized with a mean of 100 and a standard deviation of 15 based on age-matched reference data. Higher scores are always better.
The amount of change of the standardized score of processing speed between Base line and Week 12 | Base line and Week 12
  SDC test is measured using Cognitrax® which is powered by CNS Vital Signs®, a neurocognitive test system. The standardized score of processing speed is calculated from the result of this test. This score has been normalized with a mean of 100 and a standard deviation of 15 based on age-matched reference data. Higher scores are always better.
The measured value of the standardized score of executive function at Week 12 | Week 12
  SAT test is measured using Cognitrax® which is powered by CNS Vital Signs®, a neurocognitive test system. The standardized score of executive function is calculated from the result of this test. This score has been normalized with a mean of 100 and a standard deviation of 15 based on age-matched reference data. Higher scores are always better.
The amount of change of the standardized score of executive function between Base line and Week 12 | Base line and Week 12
  SAT test is measured using Cognitrax® which is powered by CNS Vital Signs®, a neurocognitive test system. The standardized score of executive function is calculated from the result of this test. This score has been normalized with a mean of 100 and a standard deviation of 15 based on age-matched reference data. Higher scores are always better.
The measured value of the standardized score of social acuity at Week 12 | Week 12
  Perception of Emotions (POET) test is measured using Cognitrax® which is powered by CNS Vital Signs®, a neurocognitive test system. The standardized score of social acuity is calculated from the result of this test. This score has been normalized with a mean of 100 and a standard deviation of 15 based on age-matched reference data. Higher scores are always better.
The amount of change of the standardized score of social acuity between Base line and Week 12 | Base line and Week 12
  POET test is measured using Cognitrax® which is powered by CNS Vital Signs®, a neurocognitive test system. The standardized score of social acuity is calculated from the result of this test. This score has been normalized with a mean of 100 and a standard deviation of 15 based on age-matched reference data. Higher scores are always better.
The measured value of the standardized score of reasoning at Week 12 | Week 12
  Non-Verbal Reasoning (NVRT) test is measured using Cognitrax® which is powered by CNS Vital Signs®, a neurocognitive test system. The standardized score of reasoning is calculated from the result of this test. This score has been normalized with a mean of 100 and a standard deviation of 15 based on age-matched reference data. Higher scores are always better.
The amount of change of the standardized score of reasoning between Base line and Week 12 | Base line and Week 12
  NVRT test is measured using Cognitrax® which is powered by CNS Vital Signs®, a neurocognitive test system. The standardized score of reasoning is calculated from the result of this test. This score has been normalized with a mean of 100 and a standard deviation of 15 based on age-matched reference data. Higher scores are always better.
The measured value of the standardized score of working memory at Week 12 | Week 12
  4-Part Continuous Performance (FPCPT) test is measured using Cognitrax® which is powered by CNS Vital Signs®, a neurocognitive test system. The standardized score of working memory is calculated from the result of this test. This score has been normalized with a mean of 100 and a standard deviation of 15 based on age-matched reference data. Higher scores are always better.
The amount of change of the standardized score of working memory between Base line and Week 12 | Base line and Week 12
  FPCPT test is measured using Cognitrax® which is powered by CNS Vital Signs®, a neurocognitive test system. The standardized score of working memory is calculated from the result of this test. This score has been normalized with a mean of 100 and a standard deviation of 15 based on age-matched reference data. Higher scores are always better.
The measured value of the standardized score of sustained attention at Week 12 | Week 12
  FPCPT test is measured using Cognitrax® which is powered by CNS Vital Signs®, a neurocognitive test system. The standardized score of sustained attention is calculated from the result of this test. This score has been normalized with a mean of 100 and a standard deviation of 15 based on age-matched reference data. Higher scores are always better.
The amount of change of the standardized score of sustained attention between Base line and Week 12 | Base line and Week 12
  FPCPT test is measured using Cognitrax® which is powered by CNS Vital Signs®, a neurocognitive test system. The standardized score of sustained attention is calculated from the result of this test. This score has been normalized with a mean of 100 and a standard deviation of 15 based on age-matched reference data. Higher scores are always better.
The measured value of the standardized score of simple attention at Week 12 | Week 12
  CPT test is measured using Cognitrax® which is powered by CNS Vital Signs®, a neurocognitive test system. The standardized score of simple attention is calculated from the result of this test. This score has been normalized with a mean of 100 and a standard deviation of 15 based on age-matched reference data. Higher scores are always better.
The amount of change of the standardized score of simple attention between Base line and Week 12 | Base line and Week 12
  CPT test is measured using Cognitrax® which is powered by CNS Vital Signs®, a neurocognitive test system. The standardized score of simple attention is calculated from the result of this test. This score has been normalized with a mean of 100 and a standard deviation of 15 based on age-matched reference data. Higher scores are always better.
The measured value of the standardized score of motor speed at Week 12 | Week 12
  FTT test is measured using Cognitrax® which is powered by CNS Vital Signs®, a neurocognitive test system. The standardized score of motor speed is calculated from the result of this test. This score has been normalized with a mean of 100 and a standard deviation of 15 based on age-matched reference data. Higher scores are always better.
The amount of change of the standardized score of motor speed between Base line and Week 12 | Base line and Week 12
  FTT test is measured using Cognitrax® which is powered by CNS Vital Signs®, a neurocognitive test system. The standardized score of motor speed is calculated from the result of this test. This score has been normalized with a mean of 100 and a standard deviation of 15 based on age-matched reference data. Higher scores are always better.

CONTACTS AND LOCATIONS:
Overall Officials: Tsuyoshi Takara, MD, Principal Investigator — Medical Corporation Seishinkai, Takara Clinic
Locations (2):
- Japan (2):
  - Nerima Medical Association Minami-machi Clinic, Nerima-ku, Tokyo
  - Medical Corporation Seishinkai, Takara Clinic, Shinagawa-ku, Tokyo

IPD SHARING:
Plan to Share IPD: No
Data sharing will be discussed among the research affiliates after the study is completed.